CLINICAL TRIAL: NCT05258760
Title: Covid Vaccine Acceptance Among Egyptian Pregnant Women
Brief Title: Covid 19 Vaccine Acceptance in Egyptian Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Other Study IDs: covid vaccine in pregnancy
Record Dates: First submitted 2022-02-25; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine vaccine acceptance and hesitancy attitudes toward coronavirus disease 2019 (COVID-19) vaccines in Egyptian pregnant women.

DETAILED DESCRIPTION:
Although 2 years passed since the Covid 19 pandemic started, no specific treatment against the disease is available. According to WHO, more than two million deaths have been recorded worldwide . Therefore, it is important to avoid infection. In the absence of an effective treatment for coronavirus disease 2019 (COVID-19) non-pharmaceutical interventions are the only available methods of disease control. Social distancing, face masks, and personal hygiene are the most effective precautions, but maintaining these actions is not practicable in the long term. As a result, vaccination becomes the most effective eradication method. (1,2) Research into development of a vaccine for SARS-CoV-2 was undertaken immediately after the disease was identified.(3) The success of a vaccine depends not only on its efficacy, but also its acceptance.

However, vaccine hesitancy has become an important threat to global health, which was pointed out by WHO in 2019.(4) Several key factors behind vaccine hesitancy include fear or mistrust of the vaccine, underestimation of the value of the vaccine, and lack of access to the vaccine.(5) Pregnant women are at increased risk of severe disease, ICU admission, and ventilation when compared with non-pregnant patients of the same age.(6-8) Therefore, pregnant women are classified as a high-risk population for COVID-19 infection.(9) Regarding this information, pregnant women have not been included in any COVID-19 vaccine clinical trials to date.(10) Even so, public health authorities, including the ACOG and the SMFM recommend that COVID-19 vaccines should be available for pregnant women if they prefer to be vaccinated.(11,12)

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at any gestational age

Exclusion Criteria:

* Covid 19 suspicious patients at time of survey.
* patients refusing survey
* obstetric emergency.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1100 pregnant women attending at kasr Alainy obstetric outpatient clinic
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-02-26 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
acceptance of and attitude toward f COVID-19 vaccination | 5 months

SECONDARY OUTCOMES:
the impact of the COVID-19 pandemic | 5 months
perception of risk related to the COVID-19 pandemic | 5 months
Improvement of vaccination status among pregnant women | 5 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hinman AR. The eradication of Polio: Have we succeeded? Vaccine. 2017 Oct 9;35(42):5519-5521. doi: 10.1016/j.vaccine.2017.09.015. Epub 2017 Sep 8. No abstract available. PMID 28890190
- [Background] Durrheim DN, Crowcroft NS, Strebel PM. Measles - The epidemiology of elimination. Vaccine. 2014 Dec 5;32(51):6880-6883. doi: 10.1016/j.vaccine.2014.10.061. Epub 2014 Nov 4. PMID 25444814
- [Background] Sharma O, Sultan AA, Ding H, Triggle CR. A Review of the Progress and Challenges of Developing a Vaccine for COVID-19. Front Immunol. 2020 Oct 14;11:585354. doi: 10.3389/fimmu.2020.585354. eCollection 2020. PMID 33163000
- [Background] 4. Volkov S, World Health Organization. Vaccine hesitancy. https:// www.who.int/news-room/ spotl ight/ten-threa ts-to- globa l-healt h-in- 2019. Accessed April 25, 2020.
- [Background] Prematunge C, Corace K, McCarthy A, Nair RC, Pugsley R, Garber G. Factors influencing pandemic influenza vaccination of healthcare workers--a systematic review. Vaccine. 2012 Jul 6;30(32):4733-43. doi: 10.1016/j.vaccine.2012.05.018. Epub 2012 May 27. PMID 22643216
- [Background] Allotey J, Stallings E, Bonet M, Yap M, Chatterjee S, Kew T, Debenham L, Llavall AC, Dixit A, Zhou D, Balaji R, Lee SI, Qiu X, Yuan M, Coomar D, Sheikh J, Lawson H, Ansari K, van Wely M, van Leeuwen E, Kostova E, Kunst H, Khalil A, Tiberi S, Brizuela V, Broutet N, Kara E, Kim CR, Thorson A, Oladapo OT, Mofenson L, Zamora J, Thangaratinam S; for PregCOV-19 Living Systematic Review Consortium. Clinical manifestations, risk factors, and maternal and perinatal outcomes of coronavirus disease 2019 in pregnancy: living systematic review and meta-analysis. BMJ. 2020 Sep 1;370:m3320. doi: 10.1136/bmj.m3320. PMID 32873575
- [Background] 7. Abdelazim IA, AbuFaza M, Al-Munaifi S. COVID-19 positive woman presented with preterm labor: case report. Gynecol Obstet Reprod Med. 2021;202:1-3.
- [Background] 8. Dey M, Singh S, Tiwari R, Nair VG, Arora D, Tiwari S. Pregnancy outcome in first 50 sars-cov- 2 positive patients at our center. Gynecol Obstet Reprod Med. 2021;202:1-6.
- [Background] 9. Control CfD, Prevention. People with certain medical conditions. Morbidity and Mortality Weekly Report CDC. 2020. https://www. cdc.gov/coron aviru s/2019-ncov/ need-extra -preca ution s/peopl e-with- medic al-condi tions.html. Accessed September 7, 2020.
- [Background] Smith DD, Pippen JL, Adesomo AA, Rood KM, Landon MB, Costantine MM. Exclusion of Pregnant Women from Clinical Trials during the Coronavirus Disease 2019 Pandemic: A Review of International Registries. Am J Perinatol. 2020 Jun;37(8):792-799. doi: 10.1055/s-0040-1712103. Epub 2020 May 19. PMID 32428965
- [Background] 11. American College of Obstetricians and Gynecologists Immunization, Infectious Disease, and Public Health Preparedness Expert Work Group in collaboration with Riley LE, Beigi R, Jamieson DJ, et al. Vaccinating pregnant and lactating patients against COVID-19. https://www.acog.org/clini cal/clini cal-guida nce/pract ice-advis ory/artic les/2020/12/vacci natin g-pregn ant-and- lacta ting-patie nts-again st-covid -19. Accessed April 25, 2020
- [Background] 12. Society for Maternal-Fetal Medicine. Society for Maternal-Fetal Medicine (SMFM) statement: SARS-CoV- 2 vaccination in pregnancy. https://s3.amazo naws.com/cdn.smfm.org/media/ 2591/SMFM_ Vacci ne_State ment_12-1- 20_( final ).pdf. Accessed April 25, 2020.